CLINICAL TRIAL: NCT02854254
Title: Peripherally Inserted Central Catheters (PICC) Reduce Phlebitis Incidence in Heart Failure Patients Receiving Prolonged Intravenous Inotropic Infusion: a Randomized Trial.
Brief Title: Peripherally Inserted Central Catheter Use for Dobutamine Infusion in Heart Failure Patients
Acronym: DOBUTAPICC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Marcelo Eidi Ochiai, Dr., InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INCOR /2012
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Congestive Heart Failure
Keywords: phlebitis; catheter; congestive heart failure; dobutamine
MeSH Terms: conditions — Heart Failure; Phlebitis | interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PICC (Experimental): peripherally inserted central catheter
  Interventions: Device: peripherally inserted central catheter
- Control (Other): peripherally venous access
  Interventions: Device: peripherally venous access

INTERVENTIONS:
Device: peripherally inserted central catheter — peripherally inserted central catheter
  Arms: PICC
Device: peripherally venous access — standard over-the-needle intravenous catheter
  Arms: Control

SUMMARY:
In decompensation of heart failure, it may occur low cardiac output. For patients in this situation, the use of inotropic may be necessary. Prolonged intravenous infusion of inotropic agents can lead to phlebitis in peripherally venous access. On the other hand, central venous access presents complications inherent in the procedure. The peripherally inserted central catheter (PICC) may be an option in this situation. The present research project is a randomized clinical trial to evaluate the incidence of phlebitis by using the PICC in comparison to the peripheral venous access. The criteria for inclusion are: advanced congestive heart failure, in use of intravenous inotropic; platelets > 50.000 mm3 and left ventricular ejection fraction (LVEF) < 0.45. Patients will be randomized to receive the PICC or keep the peripheral venous access. The main outcome will be the occurrence of phlebitis. The sample size will be of 40 patients for each group (PICC and control). The data will be analyzed by logistic regression. Will be considered significant P 0.05.

DETAILED DESCRIPTION:
Study design To evaluate the incidence of phlebitis using the PICC compared to peripheral venous access a randomized clinical trial was conducted in the period between 12/07/2012 and 10/02/2014, in adult cardiology department of a university hospital in Brazil. Patients were randomized into two groups permuted blocks of four. The sequence of randomization was built with random allocation blocks 4 through of random number tables. (3).The primary endpoint was occurrence of phlebitis.

Population Patients who were admitted with congestive heart failure of decompensated in use of intravenous inotropic agents were screened for eligibility to participate in this study. Inclusion criteria were: advanced congestive heart failure, use of vasoactive drugs, patients with platelet ≥50.000 mm3, left ventricular ejection fraction <0.45, upper limb venous system able for catheter insertion and central catheter peripherally inserted. Exclusion criteria were age <18, cardiac pacemaker or defibrillator, active systemic infection without treatment or without control, platelets <50.000 mm3, injury skin in cubital region and presence of central catheter.

Sample size calculation Based on pilot study data, we estimated the occurrence of phlebitis 20% in PICC group and 80% in control group. Considering statistical power of 80% and α-error in 5%, the sample size was estimated by 39 patients in each group. For more conservative estimation we defined 40 patients in each group (80 patients in total).Considering these values the sample size was 39 patients in each group in a more conservative estimate set the size in 40 patients for each group and 60% in the control group and 20% in the PICC group. In total 172 patients were evaluated, of these 86 patients did not meet the inclusion criteria and six did not agree to participate.

Ethics considerations Eligible patients were invited to participate and receive written information about the study objectives and procedures. After detailed explanations about the study if the patient agreed to participate they signed the informed consent. The study protocol was approved by the local ethics committee, and the study is in accordance with the principles set out in the Declaration of Helsinki. (1989) Intervention and endpoints Patients were divided into two groups: PICC Group and Control Group - peripheral venous access. In patients PICC group the catheter was inserted by the researcher and used to puncture technique guided by ultrasound (2). In the control group, patients were maintained with venous access by peripheral vein with flexible peripheral intravenous device and evaluation similar to the PICC group. The researcher evaluated daily the insertion site and asked the patient whether feel pain or not. The degree of phlebitis considered according to phlebitis scale Infusion Nurses Society (Table 1). Daily photo of all catheters and insertion site were performed. The patients were followed up to present the outcome, phlebitis; in his absence they were followed for ten consecutive days.

The dobutamine infusion was prescribed by responsible cardiologists well as the remaining drug therapy.

Statistical Analysis Categorical variables were expressed as number and percentage and compared between groups using the chi-square test (א 2) or Fisher's exact test. Continuous variables were expressed as mean, standard deviation and variance and compared between groups by Student's t test. Kaplan-Meir free-event curve (4) was built according the groups. Logistic regression analysis examined the predictive value of PICC Group and other variables for the occurrence of phlebitis, determining the odds ratio and its 95% confidence interval. Was considered statistically significant P <0.05. The primary analysis respected the principle of intention to treat, including only randomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced congestive heart failure
* In use of intravenous inotropic
* Platelets > 50.000 mm3
* Left ventricular ejection fraction < 0.45

Exclusion Criteria:

* Cardiac pacemaker or implantable defibrillator
* Active uncontrolled systemic infection
* Skin disease, central venous catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
phlebitis by visual infusion phlebitis scale (Infusion Nurses Society) | 10 days
  clinically diagnosed phlebitis by visual infusion phlebitis scale (Infusion Nurses Society) with photographic register

CONTACTS AND LOCATIONS:
Overall Officials: Antonio CP Barretto, Ph.D., Study Director — Heart Institute (InCor), University of São Paulo
Locations (1):
- Heart Institute (InCor), University of São Paulo, São Paulo, São Paulo, Brazil